CLINICAL TRIAL: NCT00205595
Title: The Distribution and Quantification of Specific Binding of the Positron Emission Tomography Tracer R)-[11C]PK11195 in Normal Human Subjects
Brief Title: Normal Binding of R-[11C]PK11195 in Human Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001/001; no other ID's
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Normal Aging
Keywords: microglia; PET; PK11195
MeSH Terms: interventions — Positron-Emission Tomography

INTERVENTIONS:
Device: Positron Emission Tomography

SUMMARY:
This is a study using Positron Emission Tomography (PET) to study the normal distribution of the PET ligand (R)-[11C]PK11195. This ligand will be used to study inflammation in the brain in several brain disorders like Alzheimer's disease and traumatic brain injury.

DETAILED DESCRIPTION:
At the University Hospital Vrije Universiteit the PET ligand PK11195 labeled with carbon-11, (R)-[11C]PK11195, will be used to study microglia activation in-vivo in patients with traumatic brain damage, Alzheimer disease, multiple sclerosis and neuritis optica, disorders with unknown pathophysiology and treatment difficulties.

PK11195 (1-(2-chlorophenyl)-N-methyl-N-1(1-methylpropyl)-3 isoquinolinecarboxamide) is a highly specific ligand for the peripheral benzodiazepine-binding site, which is particularly abundant on cells of the mononuclear macrophage line (Myers et al., 1991). In normal human brain, the peripheral-type benzodiazepine receptor ligand PK11195 exhibits low to minimal binding primarily associated with the choroid plexus, ependymal linings and glial cells. However, following neuronal damage, the cells involved in the ensuing gliosis, microglia, show a marked increase in expression of these sites (Stephenson et al., 1995;Conway et al., 1998).

PK11195 labeled with carbon-11 is a PET ligand to peripheral type benzodiazepine receptors which has already been used in patients with stroke (Ramsay et al., 1992), Rasmussen's encephalitis (Banati et al., 1999), multiple sclerosis (Banati et al., 1997) and facial nerve lesions (Myers et al., 1999). However, no tracer kinetic model for quantification has been fully validated for(R)-[11C]PK11195. In order to use (R)-[11C]PK11195 for PET-imaging of microglia activation and to use it in the longitudinal monitoring of disease progression, baseline levels of ligand uptake in a healthy control population are required. This study aims to measure (R)-[11C]PK11195 uptake in normal brain in different age groups and to develop methods for quantification of specific binding of (R)-[11C]PK11195. Because (R)-[11C]PK11195 uptake depends on regional bloodflow, each (R)-[11C]PK11195 scan will be preceded by a cerebral bloodflow scan with H215O.

OBJECTIVES

* Determine the distribution of (R)-[11C]PK11195 in normal brain
* Develop methods for quantification of specific binding of (R)-[11C]PK11195
* Determine the metabolic profile of (R)-[11C]PK11195 in healthy volunteers

DESIGN OF THE STUDY Forty healthy subjects will be recruited, 20 males and 20 females. This is an open study. The study consists of one PET scan, which will be performed at the Department of Nuclear Medicine & PET research of the VU University Medical Centre.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Good physical and mental Health which will be evaluated with medical history, a physical examination and screening laboratory tests (see appendix 1).
* Age between 18 and 40 years (20 subjects) and between 40 and 80 years (20 subjects).
* Mini Mental State score >27
* Body Mass Index (B.M.I.) between 20 -25.
* Written informed consent of the subject.
* Hb must be >8 mmol \ liter at the time of the screening.

Exclusion Criteria:

* Previous neurotrauma with loss of consciousness
* Any clinical significant abnormality of any clinical laboratory test, including drug screening, or ECG abnormality.
* History of hypertension
* Any subject who has received any investigational medication within 30 days prior to the start of this study, or who is scheduled to receive an investigational drug.
* History of psychiatric or neurological illness
* History of psychiatric or neurological illness in first-degree relatives
* History of alcohol and/or drug abuse (DSM-IV criteria)
* Current use of any medication
* Blood donation within 3 months before the scan day
* Claustrophobia
* Metal objects in or around the body (braces, pacemaker, metal fragments);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-02; Study Completion 2007-01

PRIMARY OUTCOMES:
specific binding of tracer depending on age

SECONDARY OUTCOMES:
tracer kinetic method

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Berckel, MD; PhD, Principal Investigator — VUmc Medical Centre
Locations (1):
- VU University Medical Centre, Amsterdam, Netherlands